CLINICAL TRIAL: NCT03781752
Title: Carboxylesterase 1 Genetic Variation and Methylphenidate in ADHD
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); University of Florida (Other); Children's Hospital Medical Center, Cincinnati (Other); Seattle Children's Hospital (Other)
Responsible Party: Principal Investigator, Jeffrey Newcorn, Professor, Icahn School of Medicine at Mount Sinai
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: GCO 17-0281; 1R01HD093612-01A1 (NIH)
Record Dates: First submitted 2018-12-18; First posted 2018-12-20 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: ADHD; Attention Deficit Hyperactivity Disorder
Keywords: PK Study; PD Study; Pharmacokinetics; Pharmacodynamics; Methylphenidate; MPH
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Methylphenidate; 5,10-dihydro-5-methylphenazine

STUDY DESIGN:
Intervention Model Description: The study team is performing a pharmacokinetic (PK) study using a single dose of methylphenidate (MPH) for children with ADHD diagnoses.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Methylphenidate (Experimental): Youth with ADHD
  Interventions: Drug: Methylphenidate

INTERVENTIONS:
Drug: Methylphenidate — study to determine dose
  Other Names: d,l-methylphenidate; MPH

SUMMARY:
The study team will determine the association between d,l-methylphenidate (MPH) therapeutic outcomes in ADHD patients and genetic variants of CES1 and reveal key associations between CES1 genotypes and the PK and PD of MPH.

DETAILED DESCRIPTION:
Psychostimulants are the first-line pharmacotherapy for Attention deficit-hyperactivity disorder (ADHD), and MPH accounts for approximately 50% of all stimulant usage. There has been an ~10-fold increase in MPH prescribing since 1990, with 18 million prescriptions dispensed in 2010, including 1.9 million new starts on MPH, making it the 5th most commonly prescribed medication to children ages 2 -11 and the single most frequently prescribed medication of any type in those aged 12-17 years. The annual exposure of pediatric patients to MPH is extremely high and MPH is among the most commonly prescribed chronic use oral medications for US children. Despite nearly 60 years of accrued clinical experience with MPH, the significant inter-individual variability in MPH pharmacokinetics (PK), pharmacodynamics (PD) and adverse effects is inadequately explained and unpredictable. Up to 35% of ADHD patients do not respond satisfactorily to MPH therapy, and an even larger percentage discontinues treatment despite persistent ADHD. During clinical trials of MPH in treatment-naïve patients, a significant number suffer from adverse effects that are severe and persistent enough to require dose decreases or even study withdrawal. Moreover, some severe adverse drug reactions (ADRs) - including sudden cardiac death - have been associated with MPH, although the precise reasons for these associations remain elusive and controversial. Research efforts have been made to identify genetic biomarkers associated with MPH therapeutic outcomes, almost exclusively focusing on genes related to MPH PD (e.g., dopamine transporter gene [DAT1, SLC6A3]). Unfortunately, findings from these studies have been somewhat inconsistent, equivocal or even contradictory, and they do not explain the variability in the PK of MPH. Pharmacogenomic studies in MPH-treated children have not assessed the influence of genes associated with individual variability in PK in relation to clinical response. Carboxylesterase-1 (CES1), an abundant hepatic enzyme encoded by the polymorphic CES1 gene, is the sole hepatic enzyme catalyzing the metabolism (i.e., hydrolytic deactivation) of MPH. CES1 expression and activity are known to vary substantially among individuals. The first clinically significant CES1 variant G143E (rs71647871), discovered in the study team's lab during the course of a healthy volunteer MPH PK study, led to gross impairments in MPH metabolism. This variant has been unequivocally shown in vitro and in clinical studies to lead to significantly impaired metabolism of MPH and other known CES1 substrates. The study team has established the minor allele frequency (MAF) of the G143E variant as 3-4% in the general population. Accordingly, with ~1.9 million new starts of MPH annually, an estimated 133,000 pediatric patients (i.e. G143E carrier's frequency 6-8%) with a genetically impaired ability to metabolize/deactivate the drug will receive it - exposing them to high systemic concentrations of MPH and any attendant risks or toxicities. In addition, the study team's in vitro studies have revealed that another common CES1 variant D203E (rs2307227) exhibited significantly impaired activity on MPH metabolism, although the effects on D203E on clinical response are in need of further elucidation. Furthermore, despite recent intensive research on CES1 pharmacogenetics, the functions of a large number of additional CES1 variants remain undetermined.

The study team's hypothesis is that the CES1 variants, such as the G143E and D203E, can significantly alter the expression and/or activity of CES1, thereby influencing the metabolism and disposition of MPH. These influences will be directly investigated in relation to MPH therapeutic response and tolerability in ADHD patients.

ELIGIBILITY:
Inclusion Criteria:

- Youth ages 6-17 years with ADHD as a primary diagnosis

Exclusion Criteria:

* Participants that do not have ADHD as a primary diagnosis
* Participants that do not want, require, or are not healthy enough for a single dose trial of MPH for ADHD per the clinical judgment of the treating and study clinicians
* Participants that are smokers or, are pregnant

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 500 (Estimated)
Dates: Start 2018-03-04 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Maximum methylphenidate plasma concentration (Cmax), | up to 8 Hours
  The maximum plasma concentration achieved after dosing.

SECONDARY OUTCOMES:
Time to maximum concentration (Tmax) | up 8 hours
  The time after administration of a drug when the maximum plasma concentration is reached; when the rate of absorption equals the rate of elimination.
Area under the plasma concentration curve (AUClast) | up to 8 hours
  Area under the plasma concentration-time curve from time zero to the last measurable concentration.
Area under the plasma concentration curve (AUCinf) | up to 8 hours
  Area under the plasma concentration-time curve from time zero to infinity.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Newcorn, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai; Mark Stein, PhD, Principal Investigator — University of Washington; Tanya Froehlich, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (4):
- United States (4):
  - University of Florida, Gainesville, Florida
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Seattle Children's Hospital, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhang Q, Melchert PW, Awad A, McCurdy CR, Krone B, Newcorn J, Froehlich TE, Stein MA, Raeuscher J, Zhu HJ, Markowitz JS. Increased Plasma Concentrations of 6-oxo-Methylphenidate in CES1 G134E Carriers Following a Single Oral Dose of Methylphenidate. Med Chem Res. 2025 Nov;34(11):2318-2327. doi: 10.1007/s00044-025-03477-3. Epub 2025 Oct 2. PMID 41567292